CLINICAL TRIAL: NCT00046527
Title: A Controlled, Randomized, Phase III, Multicenter, Open Label Study of ABI-007(a Cremophor Free, Protein Stabilized, Nanoparticle Paclitaxel) and Taxol in Patients With Metastatic Breast Cancer
Brief Title: Study of ABI-007 and Taxol in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA012-0
Record Dates: First submitted 2002-09-30; First posted 2002-10-03 (Estimated); Last update posted 2006-07-13 (Estimated); Status verified 2004-10

CONDITIONS: Breast Neoplasms; Metastases, Neoplasm
Keywords: Metastatic breast cancer; Taxol; Taxane
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: ABI-007

SUMMARY:
Paclitaxel (Taxol, Bristol-Meyers Squibb) has been shown to be very effective against metastatic breast cancer, as well as other cancers. Because the Taxol formulation of paclitaxel is dissolved in Cremophor, an organic solvent containing castor oil, and ethanol, prolonged intravenous administration times are required; and because the solvent has caused hypersensitivity reactions, a premedication schedule is required. ABI-007 is a new anticancer medication containing the same active ingredient as Taxol, paclitaxel, but formulated as a protein-stabilized material that is suspended in salt water and administered intravenously. The time of administration is reduced, the dose of paclitaxel can be higher than is safe for Taxol, and there is no premedication required.

This study will determine the efficacy of this new formulation of paclitaxel, as compared to Taxol, for patients with metastatic breast cancer.

This is an open label comparative study, so patients will be randomly assigned to receive either the Taxol or ABI-007 forms of paclitaxel, but will know what medication they are receiving. Treatment will be repeated every three weeks unless adverse events or treatment failure require discontinuing study medication.

DETAILED DESCRIPTION:
Taxol (Bristol-Meyers Squibb) is active against carcinomas of the ovary, breast, lung, esophagus and head and neck. A number of dose schedules of Taxol have been tested in breast cancer. Initial trials used 250 mg/m2 as a continuous infusion over 24 hours. Subsequently, shorter infusions of Taxol over three hours were tested at a dose of 175 mg/m2, with response rates of 30%-40%. Phase II studies using higher doses of Taxol at 200-250 mg/m2 had a response rate of 56% in metastatic breast cancer patients. However, at these doses, significant toxicities occurred, including neuropathy. There was a median granulocyte count nadir at 100-200 cells/mm3 for the majority of courses administered. There were also significant side effects associated with hypersensitivity to the Taxol vehicle, Cremophor-EL. These hypersensitivity reactions require a premedication schedule that includes a corticosteroid, an H2 antagonist and an antihistamine.

Abraxis BioScience is testing a reformulated form of paclitaxel without Cremophor. This formulation is a protein-stabilized, nanoparticle suspension of paclitaxel and human serum albumin in normal saline. The potential advantages of this formulation are:

* Higher tolerated doses, with greater efficacy
* Longer drug persistence in tumor as a result of the nanoparticle formulation
* Reduced infusion time
* Reduced risk of hypersensitivity with no required premedication schedule
* More rapid distribution of paclitaxel to the tissues based on pharmacokinetic data

This study will evaluate ABI-007, as compared to Taxol, in patients with metastatic breast cancer.

ELIGIBILITY:
Patients will be eligible for this trial if:

* Female, non-pregnant, non-lactating, and, if of child-bearing potential, have a negative serum pregnancy test, and use approved contraception
* Sixteen years of age or older
* Histologically or cytologically confirmed breast cancer (stage III or IV) with evidence of inoperable local recurrence or metastasis, with measurable disease
* If patient has received taxane therapy as an adjuvant he/she has not relapsed within one year of completing adjuvant taxane
* No other malignancy present within the past 5 years, except non-melanoma skin cancer, cervical intraepithelial neoplasia or in-situ cervical cancer
* Suitable candidate for paclitaxel therapy
* Hematology levels at baseline of: absolute neutrophil count of at least 1500 cells/mm3; platelet count of at least 100,000 cells/mm3; hemoglobin of at least 9 g/dL
* Chemistry levels at baseline of: AST and ALT of less than or equal to 2.5 x the upper limit of normal, if no evidence of liver metastasis; total bilirubin of less than or equal to 1.5 mg/dL; creatinine of less than or equal to 2 mg/dL; alkaline phosphatase of less than or equal to 5 x the upper limit of normal, unless there is bone metastasis but not liver metastasis
* Expected survival of at least 12 weeks
* Patient or his/her representative has signed an informed consent form

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 460
Dates: Start 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Hawkins, M.D., Study Director — Celgene Corporation
Locations (1):
- Abraxis Bioscience, Inc, Durham, North Carolina, United States